CLINICAL TRIAL: NCT01226602
Title: A Randomized, Double-blind, Placebo Controlled, Crossover, Single Centre Phase I Study to Assess the Effect of Ticagrelor on Adenosine-induced Coronary Blood Flow Velocity in Healthy Male Subjects
Brief Title: Study to Assess the Effect of Ticagrelor on Coronary Blood Flow in Healthy Male Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D5130C00067; 2010-021820-91 (EudraCT Number)
Record Dates: First submitted 2010-10-21; First posted 2010-10-22 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Blood Flow Speed; Coronary Flow Velocity
Keywords: Ticagrelor; Healthy; Coronary flow velocity; Adenosine
MeSH Terms: interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Adenosinladder; Ticagrelor (180 mg), Adenosinladder ; Theophylline (5 mg/kg), Adenosinladder
  Interventions: Drug: AZD6140
- 2 (Placebo Comparator): Adenosinladder; Placebo, Adenosinladder; Theophylline (5 mg/kg), Adenosinladder
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD6140 — P2Y12 receptor antagonist
  Other Names: Ticagrelor
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine if Ticagrelor increases the Adenosin induced coronary blood flow velocity.

ELIGIBILITY:
Inclusion Criteria:

* Suitable for ECG recording of CBFV and have no adverse reaction to adenosine challenge
* Have a body mass index between 18 and 30 kg/m2

Exclusion Criteria:

* History of clinically significant disease or disorder.
* Abnormal vital signs

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2010-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Assess the effect of Ticagrelor compared to placebo on the adenosine induced coronary blood flow velocity response by estimating the change in area under the adenosine dose response curve before and after study drug. | During 6 h at visit 2
Assess the effect of Ticagrelor compared to placebo on the adenosine induced coronary blood flow velocity response by estimating the change in area under the adenosine dose response curve before and after study drug. | During 6 h at visit 3

SECONDARY OUTCOMES:
Effect of Ticagrelor compared to placebo on the adenosine induced coronary blood flow velocity by estimating the change in area under the adenosine dose response curve before and after infusion of theophylline. | During 6 h at visit 2
Difference in basal blood flow (in the absence of adenosine) between Ticagrelor and placebo conditions before and after infusion of theophylline. | During 6h at visit 2
Difference in basal blood flow (in the absence of adenosine) between Ticagrelor and placebo conditions before and after infusion of theophylline. | During 6 h at visit 3

CONTACTS AND LOCATIONS:
Overall Officials: Jay Horrow, MD, Study Director — AstraZeneca; Marianne Hartford, MD, Principal Investigator — CTC, Göteborg; Mirjana Kujacic, MD PhD, Study Chair — AstraZeneca, Mölndal Sweden
Locations (1):
- Research Site, Uppsala, Sweden

REFERENCES:
- [Derived] Wittfeldt A, Emanuelsson H, Brandrup-Wognsen G, van Giezen JJ, Jonasson J, Nylander S, Gan LM. Ticagrelor enhances adenosine-induced coronary vasodilatory responses in humans. J Am Coll Cardiol. 2013 Feb 19;61(7):723-7. doi: 10.1016/j.jacc.2012.11.032. Epub 2013 Jan 9. PMID 23312702